CLINICAL TRIAL: NCT06029946
Title: Comparative Study of B-mode Ultrasound, Sono-Elastography, and Diffusion-weighted Imaging MRI in the Characterization of Thyroid Nodules
Brief Title: B-mode Ultrasound, Sono-Elastography, and Diffusion-weighted Imaging MRI in Thyroid Nodules
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Salma Ahmed Ragheb, assistant lecturer, Luxor university, Assiut University
Other Study IDs: Elastography and DWI thyroid
Record Dates: First submitted 2023-01-23; First posted 2023-09-08 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Thyroid Nodule
Keywords: Elastography; DWI thyroid; Thyroid Ultrasound
MeSH Terms: conditions — Thyroid Nodule | interventions — Elasticity Imaging Techniques; Ultrasonography; Magnetic Resonance Imaging; Biopsy, Fine-Needle

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: elastography, ultrasound — First local anesthesia with lidocaine 2%, then 3 smears will be obtained for each nodule using a 20-22 gauge needle, multiple passes within the lesion will be made to obtain sufficient cells, the aspirate will be spread over a glass, fixed with ethanol 95% and submitted to the pathology department to be reported.
  Other Names: MRI and fine needle biopsy

SUMMARY:
To compare the accuracy of the conventional Ultrasound 'TI-RADS', US elastography, DWI MRI, and its ADC value in characterization and differentiation of thyroid nodules.

DETAILED DESCRIPTION:
Thyroid nodules are one of the most common endocrine carcinomata (1) Most thyroid tumors have a good prognosis if early diagnosis and timely treated (2) An Ultrasound (US) exam is a safe, non-invasive imaging technique for detecting thyroid nodules (3) However, still there are no dependable criteria to discriminate malignant from benign lesions. (4) In 2009, Horvath et al proposed the Thyroid Imaging Report and Data System (TI-RADS). The new version of TI-RADS was launched by ACR in 2017. (5) Color Doppler ultrasound is also used to differentiate benign from malignant thyroid nodules. The presence of intra-nodular vascularity (Type 1b) was considered close to be malignant (6) US elastography is a novel tool to increase the diagnostic value of Ultrasound and as an adjuvant tool (7) Shear wave elastography evaluates elasticity through the propagation speed of shear waves, with the wave speed being faster in hard tissue (8) Conventional T1-and T2-weighted MR imaging can-not differentiate benign from malignant nodules (9) Diffusion-weighted imaging (DWI) is a non-invasive tool used to distinguish benign from malignant nodules (10). Malignant thyroid nodules usually have a lower ADC value attributed to cellular density and tissue perfusion. (11) Combining subjective MRI features with a quantitative measurement could improve the diagnostic yield of DW-MRI (12) The cytological examination by fine-needle aspiration (FNA) has become a reliable tool to diagnose thyroid cancers (2) Suspicious cytological findings reach up to 30% of all aspirated nodules, suggesting the need for less invasive methods (13)

ELIGIBILITY:
Inclusion Criteria:

* Patients should have a normal bleeding profile.
* Presence of solitary or multiple nodules in the thyroid gland.
* In the case of patients having multiple nodules, the nodule having suspicious ultrasound features (having TI-RADS score 4 or 5) was selected for further analysis.
* The nodules were either solid or mixed (containing both solid and cystic parts) with a predominant solid component

Exclusion Criteria:

* Contraindicated biopsy (as thrombocytopenia or bleeding disorder).
* Patient with cystic and mainly cystic nodules (TI-RADS 1 nodules).
* Nodules with complete shell-calcification which may cause color mapping artifacts.
* MRI contraindications such as Claustrophobia, MR-incompatible pacemakers, and MR-incompatible prosthetic heart valves.
* Patients with recurrent thyroid masses.
* History of operative procedure, chemo, or radiotherapy on the thyroid gland.
* Declined consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study will include patients referred to the radiology department at Assuit university presented with clinically thyroid-related neck swelling
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
compare findings of ultrasound, elastography values , ADC value with the gold standard (biopsy results) | 1 year
  To assess concordance of US suspicious features, US elastography results , MRI DWI, ADC value results, and the gold standard US-guided FNAB and ability to differentiate benign from malignant thyroid nodules.

SECONDARY OUTCOMES:
Apply ADC value Cut-off level to differentiate benign from malignant thyroid nodules | 1 year
  compare ADC value of benign and malignant nodules to obtain a cutoff level
Apply US shear elastography parameters Cut-off levels to differentiate benign from malignant thyroid nodules. | 1 year
  compare also benign and malignant nodules qualitative and quantitative elastography results.
  qualitative measurement is defined as :each nodule was assigned an elasticity score based on the color pattern type according to the classification proposed by Ueno classification method (color coded map) ranging from blue to green colors. hard nodules on the map appears as blue color and soft nodules appears as red color.
  Quantitative assessment of the velocity of US wave propagation through tissue. measurement units are: kilopascal (Kpa), and shear wave velocity (m/sec).
Compare individual specific US features with the Gold standard US-guided FNAB which is more important. | 1 year
  which is the most suspicious feature in ulrasound.
  The five Ultrasound suspicious features are:
  1. predominantly Solid nodule.
  2. Marked hypoechogenicity.
  3. Microlobulated or irregular margins.
  4. Micro-Calcifications.
  5. Taller-than-wide in shape with a ratio ≥ 1.
Study role of color doppler in differentiating benign from malignant thyroid nodules | 1 year
  which pattern of color doppler study is the most suspicious:
  Classified into 4 groups:
  0= Avascular.
  1a= Peri-nodular vascularity.
  1b= Intra-nodular vascularity.
  1c= Peri-nodular and intranodular vascularity.
Compare the added value of combining different modalities, which have the higher sensitivity and specificity in differentiating benign from malignant thyroid nodules | 1 year
  combination of different imaging modalities which will have the best sensitivity and specificity for diagnosis of malignant thyroid nodules

CONTACTS AND LOCATIONS:
Overall Officials: noha mohamed ali, assistant professor, Study Chair — nohamohamedali@yahoo.com; sami Abdel_Aziz Khalil, professor, Study Director — samyKhalil24@gmail.com

REFERENCES:
- [Result] Qin P, Wu K, Hu Y, Zeng J, Chai X. Diagnosis of Benign and Malignant Thyroid Nodules Using Combined Conventional Ultrasound and Ultrasound Elasticity Imaging. IEEE J Biomed Health Inform. 2020 Apr;24(4):1028-1036. doi: 10.1109/JBHI.2019.2950994. Epub 2019 Nov 4. PMID 31689223
- [Result] Wu Q, Li Y, Liu Y, Shen J, Wang Y, Yi X, Hu B. The value of conventional sonography and ultrasound elastography in decision-making for thyroid nodules in different categories of the Bethesda system for reporting thyroid cytopathology. Clin Hemorheol Microcirc. 2020;74(3):255-266. doi: 10.3233/CH-180533. PMID 31683465
- [Result] Floridi C, Cellina M, Buccimazza G, Arrichiello A, Sacrini A, Arrigoni F, Pompili G, Barile A, Carrafiello G. Ultrasound imaging classifications of thyroid nodules for malignancy risk stratification and clinical management: state of the art. Gland Surg. 2019 Sep;8(Suppl 3):S233-S244. doi: 10.21037/gs.2019.07.01. PMID 31559190
- [Result] Zhang WB, Li JJ, Chen XY, He BL, Shen RH, Liu H, Chen J, He XF. SWE combined with ACR TI-RADS categories for malignancy risk stratification of thyroid nodules with indeterminate FNA cytology. Clin Hemorheol Microcirc. 2020;76(3):381-390. doi: 10.3233/CH-200893. PMID 32675401
- [Result] Swan KZ, Bonnema SJ, Jespersen ML, Nielsen VE. Reappraisal of shear wave elastography as a diagnostic tool for identifying thyroid carcinoma. Endocr Connect. 2019 Aug;8(8):1195-1205. doi: 10.1530/EC-19-0324. PMID 31340198
- [Result] Kwak JY, Kim EK. Ultrasound elastography for thyroid nodules: recent advances. Ultrasonography. 2014 Apr;33(2):75-82. doi: 10.14366/usg.13025. Epub 2014 Feb 26. PMID 24936499
- [Result] Wang H, Wei R, Liu W, Chen Y, Song B. Diagnostic efficacy of multiple MRI parameters in differentiating benign vs. malignant thyroid nodules. BMC Med Imaging. 2018 Dec 3;18(1):50. doi: 10.1186/s12880-018-0294-0. PMID 30509198
- [Result] Gorgulu FF. Which Is the Best Reference Tissue for Strain Elastography in Predicting Malignancy in Thyroid Nodules, the Sternocleidomastoid Muscle or the Thyroid Parenchyma? J Ultrasound Med. 2019 Nov;38(11):3053-3064. doi: 10.1002/jum.15013. Epub 2019 Apr 29. PMID 31037753
- [Result] Cantisani V, David E, Grazhdani H, Rubini A, Radzina M, Dietrich CF, Durante C, Lamartina L, Grani G, Valeria A, Bosco D, Di Gioia C, Frattaroli FM, D'Andrea V, De Vito C, Fresilli D, D'Ambrosio F, Giacomelli L, Catalano C. Prospective Evaluation of Semiquantitative Strain Ratio and Quantitative 2D Ultrasound Shear Wave Elastography (SWE) in Association with TIRADS Classification for Thyroid Nodule Characterization. Ultraschall Med. 2019 Aug;40(4):495-503. doi: 10.1055/a-0853-1821. Epub 2019 May 28. PMID 31137050
- [Result] Aghaghazvini L, Maheronnaghsh R, Soltani A, Rouzrokh P, Chavoshi M. Diagnostic value of shear wave sonoelastography in differentiation of benign from malignant thyroid nodules. Eur J Radiol. 2020 May;126:108926. doi: 10.1016/j.ejrad.2020.108926. Epub 2020 Mar 3. PMID 32171916
- See also: Conventional ultrasound, color Doppler, TI-RADS, and shear wave elastography for thyroid nodule differentiation: a study of efficacy compared with the histopathology results — https://ejrnm.springeropen.com/articles/10.1186/s43055-021-00474-5#citeas
- See also: Diagnostic accuracy of B-mode ultrasound, ultrasound elastography and diffusion weighted MRI in differentiation of thyroid nodules (prospective study) — https://ejrnm.springeropen.com/articles/10.1186/s43055-021-00640-9
- See also: DIFFUSION WEIGHTED MAGNETIC RESONANCE IMAGING IN DIFFERENTIATION OF BENIGN AND MALIGNANT THYROID NODULES — https://www.medicaljournalofcairouniversity.net/index.php/2014-10-21-22-15-18/med-j-cairo-univ-vol-88-2020/116-vol-88-december-2020/4790-diffusion-weighted-magnetic-resonance-imaging-in-differentiation-of-benign-and-malignant-thyroid-nodules